CLINICAL TRIAL: NCT06390475
Title: Optimizing Diagnosis of Splanchic Vein Thrombosis With MR Direct Thrombus Imaging, the Rhea Study
Brief Title: Optimizing Diagnosis of Splanchic Vein Thrombosis With MRDTI (Rhea)
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: ISTH (Unknown); Trombosestichting Nederland (Unknown)
Responsible Party: Principal Investigator, Erik Klok, Prof. Dr., Leiden University Medical Center
Other Study IDs: P18.089
Record Dates: First submitted 2024-04-18; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Splanchnic Vein Thrombosis
Keywords: MR Direct Thrombus Imaging; Splanchnic vein thrombosis; Diagnostic management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic splanhnic thrombosis: Chronic Splanchnic vein thrombosis is defined by incident SVT with chronic thrombi on 2 serial imaging tests with an at least 3 months interval.
  Interventions: Diagnostic Test: MR Direct Thrombus Imaging (MRDTI)
- Acute splanchnic thrombosis: Acute splanchnic vein thrombosis is defined as acute symptomatic or acute incidental asymptomatic thrombosis in the mesenteric, splenic, portal or hepatic veins. Acute symptomatic thrombosis refers to acute onset (< 2 week existent) of symptoms characteristic for SVT thrombosis (including but not limited to abdominal pain) with SVT confirmed with DUS, CTA or MRA, dependent on the anatomical location. Acute incidental asymptomatic thrombosis refers to an incidentally detected SVT with DUS, CTA or MRA, absent on previous diagnostic tests performed in the last 2 weeks before the new incidental finding, in patients without symptoms characteristic of SVT.
  Interventions: Diagnostic Test: MR Direct Thrombus Imaging (MRDTI)

INTERVENTIONS:
Diagnostic Test: MR Direct Thrombus Imaging (MRDTI) — Both groups will get the same MRDTI, the study is a proof-of-concept study to investigate if MRDTI can reliable distinguish between acute and chronic splanchnic thrombosis.

SUMMARY:
The Rhea-study is a multicenter prospective diagnostic proof-of-concept study

There is an unquestionable need for improved diagnostic approaches for (incidental) SVT. The researchers plan to evaluate the MRDTI technique, that has been shown to be accurate in other settings of difficult-to-diagnosis venous thrombosis, for the notoriously challenging diagnosis of incidental SVT. This study targets an important unmet need and will provide the basis for precision medicine for patients with SVT in the near future, i.e. the possibility of assessment of the age of the thrombus in patients with incidental SVT, which is of utmost importance for determination of the indication for anticoagulant therapy.

If this hypothesis is proven true, i.e. sensitivity of MRDTI for SVT is indeed >90%, the investigators will proceed with performing a randomized controlled outcome study in which patients with possible/probable chronic SVT with normal MRDTI test results and no other indications for anticoagulant therapy. These patients will be randomized between active therapeutically dosed anticoagulation versus no anticoagulation, to compare clinical outcome with regard to the occurrence of venous thromboembolism and/or Progressive symptomatic SVT as well as major bleeding.

DETAILED DESCRIPTION:
Background:

Splanchnic vein thrombosis (SVT) is one of the manifestations of unusual site venous thromboembolism (VTE). SVT includes portal vein thrombosis (PVT), mesenteric vein hrombosis (MVT), splenic vein thrombosis (SpVT) and the Budd-Chiairi syndrome (BCS).There is no validated clinical algorithm for the diagnosis of SVT and there are no specific laboratory tests available to confirm or rule out the disease. Particularly, D-dimer tests do not have a role in the diagnosis of SVT, due to its low specificity and the high percentage of false positive results, especially in patients with cancer, liver cirrhosis or underlying inflammatory conditions, present in more than half of the total SVT population. Thus the diagnosis of SVT relies on imaging tests alone. Whereas Doppler ultrasound is the imaging test of choice for most forms of SVT, its sensitivity is only 90%, as is the sensitivity of CT angiography (CTA). MR angiography (MRA) has been reported to have 90-100% sensitivity for SVT, but this technique is limited by the need to administer a contrast agent. Furthermore, in studies evaluating the accuracy of MRA for the diagnose of SVT, gold standard for SVT (surgical validation) was lacking. Importantly, many of SVT diagnoses in clinical practice (up to 30%) are incidental findings, i.e. findings on imaging tests of the abdomen performed for another reason than suspected SVT. Whereas the diagnosis of symptomatic SVT is often challenging, the correct diagnosis of acute versus chronic SVT is even more difficult, as neither of the current available imaging tests is helpful in determination of the age and clinical relevance of the thrombus, especially in non-symptomatic patients. Due to this impossibility to determine whether the incidentally observed thrombosis is acute, chronic or even an imaging artefact, the vast majority of patients with incidental SVT are treated with often lifelong anticoagulants. It is widely acknowledged that this practice likely results in overdiagnosis and unjust exposure to anticoagulant therapy with associated risk of bleeding. An alternative imaging technique for more accurate diagnosis of SVT is MR Direct hrombus Imaging (MRDTI). This technique is in an advanced stage of development (Theia study, NCT02262052, supported by TSN grant 2013-02) and is close to implementation in clinical practice. The method is based on the formation of methemoglobin in a fresh thrombus leading to shortening of the T1 signal. It does not require contrast dye. Both the diagnostic accuracy (sensitivity 97-100%, specificity 100%) as well as the inter-observer agreement of MRDTI for first and recurrent DVT of the leg were reported to be excellent (kappa 0.89-0.98). Moreover, it was shown to accurately differentiate acute from chronic thrombosis. There is an unquestionable need for improved diagnostic approaches for (incidental) SVT. The researchers plan to evaluate the MRDTI technique, that has been shown to be accurate in other settings of difficult-to-diagnosis venous thrombosis, for the notoriously challenging diagnosis of incidental SVT. This study targets an important unmet need and will provide the basis for precision medicine for patients with SVT in the near future, i.e. the possibility of assessment of the age of the thrombus in patients with incidental SVT, which is of utmost importance for determination of the indication for anticoagulant therapy.

Study design:

This study is a prospective diagnostic proof of concept study to explore the diagnostic accuracy of MRDTI in the diagnostic management of acute and chronic SVT. This will be achieved by performing MRDTI scans to adjust and optimize the DTI scan sequence in 3-5 patients with confirmed, acute SVT. If a reproducible clearly positive DTI signal is achieved in all patients, the study can proceed with the inclusion of cohort 1 and 2, i.e. 35 patients with confirmed acute SVT and in 35 patients with confirmed, chronic SVT. All scans will be evaluated post-hoc by expert readers blinded for the final diagnosis. It is predetermined that at least five patients of each SVT site (PVT, SpVT and BCS and at least five patients of each SVT risk factor (oncologic, post-surgical and inflammatory/infectious) will be included. To make sure that cohort 1 is generally similar to cohort 2 frequency matching will be performed, in which all controls will be selected to get the same distribution according to SVT site and risk factor as cases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed acute SVT; definitions provided in paragraph 4.2 (Cases, group 1)
2. Patients with confirmed non-symptomatic chronic SVT defined by incident SVT with chronic thrombi on 2 serial imaging tests with at least 3 months interval (controls, group 2)
3. Aged 18 years and older
4. Willing and able to give informed consent

Exclusion Criteria:

1. MRI contra-indication (including but not limited to a cardiac pacemaker or subcutaneous defibrillator; vascular clips in the cerebral vessels; metal splinter in the eye, a hearing aid that cannot be removed; a neurostimulator that cannot be removed; a hydrocephalus pump)
2. A medical condition, associated illness or co-morbid circumstances that precludes completion of the study procedures (MRI and 90-day follow-up assessment), including but not limited to lifeexpectancy less than 3 months, inability to lie flat, morbid obesity preventing use of MR and claustrophobia.
3. Patients with decompensated liver disease with Child-Pugh class C cirrhosis (since MRDTI evaluation will be inadequate in these patients)
4. Patients with suspected tumour thrombus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a proven splanchnic vein thrombosis either acute or non-symptomatic chronic SVT defined by incident SVT with chronic thrombi on 2 serial imaging tests with at least 3 months interval.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Estimated)
Dates: Start 2019-03-22 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of MRDTI | This outcome will be analysed after adjudication, after the follow-up period of 3 months.
  The primary objective of this study is to explore the diagnostic accuracy of MRDTI in the diagnostic management of acute and chronic SVT in a prospective diagnostic proof of concept study.

SECONDARY OUTCOMES:
Optimizing MRDTI sequences | This outcome will be analysed immediately after the inclusion of the first 3-5 acute SVT patients.
  To optimise MRDTI sequences for imaging of SVT
Interobserver agreement | This outcome will be analysed after adjudication, after the follow-up period of 3 months.
  To assess the interobserver agreement of the readers of MRDTI for suspected SVT

CONTACTS AND LOCATIONS:
Overall Officials: F.A. Klok, Prof., Principal Investigator — Study Principal Investigator
Locations (3):
- Italy (2):
  - Gemelli Hospital, Rome
  - Varese hospital, Varese
- Erasmus Medisch Centrum, Rotterdam, Netherlands

REFERENCES:
- [Background] Riva N, Ageno W. Approach to thrombosis at unusual sites: Splanchnic and cerebral vein thrombosis. Vasc Med. 2017 Dec;22(6):529-540. doi: 10.1177/1358863X17734057. PMID 29202678
- [Background] Dai J, Qi X, Peng Y, Hou Y, Chen J, Li H, Guo X. Association between D-dimer level and portal venous system thrombosis in liver cirrhosis: a retrospective observational study. Int J Clin Exp Med. 2015 Sep 15;8(9):15296-301. eCollection 2015. PMID 26629017
- [Background] Riva N, Ageno W. Clinical manifestations and imaging tools in the diagnosis of splanchnic and cerebral vein thromboses. Thromb Res. 2018 Mar;163:252-259. doi: 10.1016/j.thromres.2017.06.030. Epub 2017 Jun 27. PMID 28673473
- [Background] Cakmak O, Elmas N, Tamsel S, Demirpolat G, Sever A, Altunel E, Killi R. Role of contrast-enhanced 3D magnetic resonance portography in evaluating portal venous system compared with color Doppler ultrasonography. Abdom Imaging. 2008 Jan-Feb;33(1):65-71. doi: 10.1007/s00261-007-9229-x. PMID 17440768
- [Background] Kreft B, Strunk H, Flacke S, Wolff M, Conrad R, Gieseke J, Pauleit D, Bachmann R, Hirner A, Schild HH. Detection of thrombosis in the portal venous system: comparison of contrast-enhanced MR angiography with intraarterial digital subtraction angiography. Radiology. 2000 Jul;216(1):86-92. doi: 10.1148/radiology.216.1.r00jl2386. PMID 10887231
- [Background] Riva N, Ageno W, Schulman S, Beyer-Westendorf J, Duce R, Malato A, Santoro R, Poli D, Verhamme P, Martinelli I, Kamphuisen P, Dentali F; International Registry on Splanchnic Vein Thrombosis (IRSVT) study group. Clinical history and antithrombotic treatment of incidentally detected splanchnic vein thrombosis: a multicentre, international prospective registry. Lancet Haematol. 2016 Jun;3(6):e267-75. doi: 10.1016/S2352-3026(16)30020-5. Epub 2016 May 11. PMID 27264036

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/75/NCT06390475/Prot_SAP_000.pdf